CLINICAL TRIAL: NCT05109507
Title: Pilot Randomized Trial of Visitor Mindset: A Single-Session Self-Guided Digital Intervention Targeting Emotional Awareness, Clarity, and Acceptance Among Adults With Anxiety and/or Depression Symptoms
Brief Title: Single-Session Intervention Targeting Emotional Awareness, Clarity, and Acceptance to Reduce Depression/Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Principal Investigator, Corey Roos, Assistant Professor of Psychiatry, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2000030587
Record Dates: First submitted 2021-10-18; First posted 2021-11-05 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visitor Mindset (Experimental): Single-session, self-guided web-based intervention (~30 to 45 minutes) hosted on Qualtrics with animated videos, audio-guided exercises, graphics, text-based material, and interactive questions. The intervention is designed to enhance emotional awareness, clarity, and acceptance, as well as modify beliefs about the duration and usefulness of negative emotions.
  Interventions: Behavioral: Visitor Mindset
- Relaxing with Nature (Active Comparator): Single-session self-guided web-based intervention (~30 to 45 minutes) hosted on Qualtrics with videos (real-life images), text-based material, and questions. There are five videos showing different types of nature (e.g., forest scenes, beach scenes, etc.). Each video includes a sequence of pleasant nature photos (shown about 6 seconds each) with relaxing music in the background.
  Interventions: Behavioral: Relaxing with Nature

INTERVENTIONS:
Behavioral: Visitor Mindset — Single-session, self-guided intervention
  Arms: Visitor Mindset
Behavioral: Relaxing with Nature — Single-session, self-guided intervention
  Arms: Relaxing with Nature

SUMMARY:
Two-arm, parallel group randomized clinical trial conducted via Mturk comparing a single-session web-based intervention called Visitor Mindset versus a control intervention (nature videos with relaxing music) for adults with depression and/or anxiety symptoms

DETAILED DESCRIPTION:
Procedures include completing: (1) pre-intervention assessments; (2) one of two single-session web-based intervention (approximately 30 to 45 minutes each); (3) post-intervention assessments, including survey questions following a negative affect induction (brief film clip); and (4) a 2-week follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older
* English-speaking
* At least mild anxiety and/or depression symptoms, as indicated by a score of 3 or greater on the 4-item Patient Health Questionnaire (PHQ-4)

Exclusion Criteria:

* fail to meet above-listed inclusion criteria
* exit the study prior to condition randomization
* obvious lack of English fluency in open response questions
* responding with random text in open response questions
* respond with either copy/pasted responses from text earlier in the intervention to any of free response questions
* participants with a completion time less than 180 seconds for the baseline survey assessment (taking about 1.5 seconds per question) OR who fail all three attention check questions in the baseline survey, indicating very careless, random, inattentive and/or hasty responding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 530 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in anxiety and depression symptoms | Baseline to 2-week follow-up
  Patient Health Questionnaire-Anxiety Depression Scale (PHQ-ADS). Total scores range from 0 to 27, with higher scores indicating greater anxiety/depression symptoms.

SECONDARY OUTCOMES:
Change over time in functional impairment | Baseline to 2-week follow-up
  Work and Social Adjustment Scale (WSAS). Total scores range from 0 to 40, with higher scores indicating greater functional impairment.
State emotional awareness, clarity, and acceptance following negative affect induction | Immediate post-intervention
  Adapted state version of Emotion Regulation Skills Questionnaire (ERSQ). Total scores for each subscale range from 0 to 12, with higher scores indicating greater state emotional awareness, clarity. or acceptance.
State non-acceptance of emotions | Immediate post-intervention
  Non-acceptance subscale of the State Difficulties in Emotion Regulation Scale (S-DERS). Total scores range from 0 to 12, with higher scores indicating greater state emotional non-acceptance.
Change over time in emotional awareness, clarity, and acceptance | Baseline to 2-week follow-up
  Emotion Regulation Skills Questionnaire (ERSQ). Total scores for each subscale range from 0 to 12, with higher scores indicating greater emotional awareness, clarity. or acceptance.
Change over time in non-acceptance of emotions | Baseline to 2-week follow-up
  Non-acceptance subscale of the Difficulties in Emotion Regulation Scale (DERS). Total scores range from 0 to 12, with higher scores indicating greater state emotional non-acceptance.
Change over time in beliefs about the usefulness of negative emotions | Baseline to 2-week follow-up
  Emotion Beliefs Questionnaire (EBQ). Total scores range from 0 to 16, with higher scores indicating greater beliefs that emotions are not useful or harmful
Change over time in beliefs about the duration of negative emotions | Baseline to 2-week follow-up
  duration subscale (2 items) of the Leahy Emotion Schema Scale (LESS) and 2 items ("When I'm upset, I believe that I will remain that way for a long time" and "When I'm upset, I believe that I'll end up feeling very depressed") from the modification subscale of the Difficulties in Emotion Regulation Scale (DERS). Total scores range from 0 to 16, with higher scores indicating greater maladaptive beliefs about the duration of emotions (they last will last forever)

OTHER OUTCOMES:
Change in self-compassion | Baseline to 2-week follow-up
  Self-Compassion Scale (SCS). Total scores range from 0 to 48, with higher scores indicating greater self-compassion.
Repetitive negative thinking | Baseline to 2-week follow-up
  Persistent and Intrusive Negative Thoughts Scale (PINTS). Total scores range from 0 to 20, with higher scores indicating greater repetitive negative thinking.
Avoidance | Baseline to 2-week follow-up
  Cognitive avoidance subscale of the Coping Response Inventory (CRI). Total scores range from 0 to 20, with higher scores indicating greater avoidance.
Problem-solving | Baseline to 2-week follow-up
  Problem-solving subscale of the Coping Response Inventory (CRI). Total scores range from 0 to 20, with higher scores indicating greater problem-solving.
Positive Reappraisal | Baseline to 2-week follow-up
  Positive reappraisal subscale of the Coping Response Inventory (CRI). Total scores range from 0 to 20, with higher scores indicating greater positive reappraisal.
Pain intensity | Baseline to 2-week follow-up
  Single item visual analogue scale (0 to 10) of pain intensity drawn from the Brief Pain Inventory (BPI)
Pain interference | Baseline to 2-week follow-up
  Single item visual analogue scale (0 to 10) of pain interference ("To what extent has pain interfered with your ability to enjoy life") drawn from the Brief Pain Inventory (BPI)
Pain catastrophizing | Baseline to 2-week follow-up
  Single item ("When I feel pain, it is terrible, and I feel it is never going to get any better") drawn from the Pain Catastrophizing Scale (PCS), rated on a scale from 0 to 4.
Alcohol use | Baseline to 2-week follow-up
  Daily Drinking Questionnaire (DDQ). Minimum score is 0 and maximum score is not known and depends on how many drinks the participant reports. Higher scores indicate greater alcohol use.
Alcohol craving | Baseline to 2-week follow-up
  Single item visual analogue scale (0 to 10) of craving severity
Affective self-compassion | Baseline to 2-week follow-up
  Affective Self-Compassion Questionnaire (ASCQ). Total scores range from 0 to 40, with higher scores indicating greater affective self-compassion.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale University School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roos CR, Bricker J, Kiluk B, Trull TJ, Bowen S, Witkiewitz K, Kober H. A smartphone app-based mindfulness intervention to enhance recovery from substance use disorders: Protocol for a pilot feasibility randomized controlled trial. Contemp Clin Trials Commun. 2024 Jul 26;41:101338. doi: 10.1016/j.conctc.2024.101338. eCollection 2024 Oct. PMID 39233850